CLINICAL TRIAL: NCT01775514
Title: Occurrence Rate of Non-Small Cell Lung, Colon Cancer, Breast Cancer, Gastric Cancer and Malignant Melanoma in Turkey & Diagnosis and Treatment Characteristics Turkish "Non-Small Cell Lung-Colon-Gastric-Breast (CGB) Cancer and Malignant Melanoma" Study
Brief Title: A Non-Interventional Study of the Occurrence Rate of Non-Small Cell Lung Cancer, Colon Cancer, Breast Cancer, Gastric Cancer and Malignant Melanoma in Turkey, and Diagnosis and Treatment Characteristics
Status: Completed | Type: Observational
Sponsor: Hoffmann-La Roche (Industry)
Responsible Party: Sponsor
Other Study IDs: ML28579
Record Dates: First submitted 2013-01-18; First posted 2013-01-25 (Estimated); Last update posted 2016-11-02 (Estimated); Status verified 2016-11

CONDITIONS: Cancer
MeSH Terms: conditions — Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective

GROUPS / COHORTS (1):
- Participants With Cancer: Participants from Turkey with non-small cell lung, colon cancer, breast cancer, gastric cancer and malignant melanoma will be included.

SUMMARY:
This non-interventional study will assess the occurrence rate of non-small cell lung cancer, colon cancer, breast cancer, gastric cancer and malignant melanoma in Turkey, and the diagnostic methods and treatments used. Data will be collected over 36 months.

ELIGIBILITY:
Inclusion Criteria:

* Participants diagnosed with non-small cell lung, colon, breast, gastric cancer and melanoma
* Participants who give consent to the collection of their information after the first record and pathological confirmation of their cancer

Exclusion Criteria:

* Participants not living in the city or representative region of the study center

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants with non-small cell lung cancer, colon cancer, breast cancer, gastric cancer and malignant melanoma in Turkey
Sampling Method: Probability Sample
Enrollment: 32277 (Actual)
Dates: Start 2012-10; Primary Completion 2015-10 (Actual); Study Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Number of Participants with Malignant Melanoma (Occurrence Rate), Defined as New Cases Recorded in the Relevant Region in 1 Year/Population of the Region | 36 months
Number of Participants with Non-Small Cell Lung Cancer (Occurrence Rate), Defined as New Cases Recorded in the Region in 1 Year Divided by (/) Population of the Region | 36 months
Number of Participants with Colon Cancer (Occurrence Rate), Defined as New Cases Recorded in the Relevant Region in 1 Year/Population of the Region | 36 months
Number of Participants with Breast Cancer (Occurrence Rate), Defined as New Cases Recorded in the Relevant Region in 1 Year/Population of the Region | 36 months
Number of Participants with Gastric Cancer (Occurrence Rate), Defined as New Cases Recorded in the Relevant Region in 1 Year/Population of the Region | 36 months

SECONDARY OUTCOMES:
Percentage of Participants Categorized by Tumor Size | 36 months
Percentage of Participants Categorized by Histopathology Diagnosis | 36 months
Percentage of Participants Categorized by the Staging System | 36 months
Percentage of Participants Categorized by Surgery Type | 36 months
Percentage of Participants Categorized by Type of Treatments Administered (ie, Adjuvant and Neoadjuvant Treatments) | 36 months
Percentage of Participants With Metastasis Categorized by Treatment Regimens Used (ie, First-line, Second-line, Third-line, or Forth-line Chemotherapy) | 36 months
Overall Survival (OS) | 36 months
Progression-free Survival (PFS) as Assessed by Response Evaluation Criteria in Solid Tumors (RECIST) | 36 months
Percentage of Participants With Family History of Cancer and Other Conditions | 36 months
Percentage of Participants With History of Another Primary Cancer | 36 months
Percentage of Participants Categorized by Diagnostic Methods | 36 months
Percentage of Participants With Metastasis | 36 months
Percentage of Participants Categorized by Tumor Localization | 36 months

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Trials, Study Director — Hoffmann-La Roche
Locations (19):
- Turkey (Türkiye) (19):
  - Adana
  - Afyonkarahisar
  - Ankara
  - Baıkesir
  - Bursa
  - Denizli
  - Diyarbakır
  - Edirne
  - Erzurum
  - Gaziantep
  - Isparta
  - Istanbul
  - Izmir
  - Kayseri
  - Konya
  - Malatya
  - Sıhhiye, Ankara
  - Tokat Province
  - Trabzon